CLINICAL TRIAL: NCT06978127
Title: Technology Assisted Collaborative Care Intervention (TĀCcare) 2.0 Implementation Trial to Improve Patient-centered Outcomes in Patients on Hemodialysis
Brief Title: Technology Assisted Collaborative Care Intervention to Improve Patient-centered Outcomes in Dialysis Patients
Acronym: TACcare 2 0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of New Mexico (Other)
Responsible Party: Principal Investigator, Manisha Jhamb, Associate Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24070169; 2R01DK114085-06 (NIH)
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
Keywords: Chronic Kidney Disease; Hemodialysis; Pain; Depression; Fatigue
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pain; Depression; Fatigue

STUDY DESIGN:
Intervention Model Description: The intervention is a hybrid Type II effectiveness-implementation, cluster randomized trial of TĀCcare 2.0 facilitated by dialysis staff in a real-world setting.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology Assisted Stepped Collaborative Care Group (Active Comparator): Participants in the Technology Assisted Stepped Collaborative Care group will receive a stepped-approach for pharmaco and/or Cognitive Behavioral Therapy (CBT) and individualization of treatment to improve symptoms of fatigue, pain and/or depression, in a real-world setting.
  Interventions: Behavioral: Technology Assisted Stepped Collaborative Care
- Usual Care Group (Active Comparator): Participants in the Usual Care Group will continue with their usual care.
  Interventions: Other: Usual Care Arm

INTERVENTIONS:
Behavioral: Technology Assisted Stepped Collaborative Care — The TĀCcare 2.0 intervention will provide pharmacotherapy recommendations and/or CBT for pain, fatigue and depression. A stepped-treatment approach will be used to intensify treatment. CBT will be provided through 12 weekly telehealth sessions (done during dialysis treatment or from home) with the behavioral specialist. Booster sessions will be used to enhance the maintenance of effect following the initial intervention to complete a total 12 month intervention. A collaborative care approach will be used so that patients' symptom management will be integrated with their dialysis treatment. Throughout the study, participants will be asked to complete phone surveys about their symptoms and health.
  Arms: Technology Assisted Stepped Collaborative Care Group
Other: Usual Care Arm — Participants in the Usual Care Arm will continue with their usual care.
  Arms: Usual Care Group

SUMMARY:
The goal of this study is to learn if a collaborative care intervention of pharmaco-therapy and/or cognitive behavioral therapy (CBT), delivered in a real-world setting, improves symptoms of pain, fatigue and/or depression.

DETAILED DESCRIPTION:
The goal of this study is to conduct a hybrid Type II effectiveness-implementation, cluster randomized trial of TĀCcare 2.0 facilitated by dialysis staff in a real-world setting. This is a multi-center, dialysis-clinic level cluster randomized trial of 424 patients from 36 dialysis clinics comparing TACcare 2.0 facilitated by dialysis staff versus usual care. Patients' dialysis clinic will be placed randomly into one of two study groups: the Technology Assisted Stepped Collaborative Care Intervention Group or the Usual Care Group.

The intervention will target three of the most debilitating End State Kidney Disease (ESKD) related symptoms- fatigue, pain and depression. A stepped collaborative care approach for pharmaco and/or CBT allows for shared decision-making and individualization of treatment according to a patient's clinical status, preferences and treatment response. The TĀCcare 2.0 intervention will build on successful design elements of the original intervention, enhance depression management strategies and increase durability of effect by incorporating monthly longitudinal telemedicine-delivered booster sessions to complete a total 12-month intervention. Additionally, using a collaborative care approach, the patients' symptom management will be integrated with their dialysis treatment, thus increasing patient acceptability and adherence.

ELIGIBILITY:
Eligibility Criteria:

1. age 18 years or older;
2. undergoing thrice-weekly maintenance hemodialysis (HD) for > 3 months;
3. English or Spanish speaking;
4. able to provide informed consent

Ineligibility Criteria:

1. active thought disorder, delusions or active suicidal ideation
2. active substance abuse
3. enrolled in hospice or life expectancy < 6 months (based on clinician's judgement)
4. too ill or cognitively impaired to participate based on renal provider's judgement
5. living kidney transplant scheduled in <3 months
6. undergoing active cancer treatment.
7. enrolled in another research study
8. plan to transition to home dialysis within 3 months
9. plan to move to another dialysis facility within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
TĀCcare 2.0 Effectiveness evaluation/Change in fatigue (co-primary outcome) | 6 months
  Change in fatigue is a primary outcome. The Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) will be used to measure fatigue. Scores range from 0-52 with lower scores indicating greater fatigue.
TĀCcare 2.0 Effectiveness evaluation/Change in Pain Intensity (co-primary outcome) | 6 months
  Change in pain intensity score is also a primary outcome measure. The Brief Pain Inventory (BPI) will be used to measure pain intensity. The BPI uses a scale of 0 to 10. Higher scores on the pain intensity scale indicate greater pain severity.
TĀCcare 2.0 Effectiveness evaluation/Change in Depression (co-primary outcome) | 6 months
  Change in depression severity score is also a primary outcome measure. The Beck Depression Inventory-II will be used to measure the depression severity score. Each item is scored on a 4 point scale ranging from 0 to 3, allowing for a total score ranging from 0 to 63. Higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Fatigue | 3 and 12 months
  Change in fatigue measured by The Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F). Scores range from 0-52 with lower scores indicating greater fatigue.
Pain Intensity | 3 and 12 months
  Change in pain intensity measured by Brief Pain Inventory (BPI), which uses a scale of 0 to 10. Higher scores on the pain intensity scale indicate greater pain severity.
Depression | 3 and 12 months
  Change in depression severity score using The Beck Depression Inventory-II (BDI-II). Each item is scored on a 4 point scale ranging from 0 to 3, allowing for a total score ranging from 0 to 63. Higher scores indicate more severe symptoms.
Pain interference | 3, 6 and 12 months
  Brief Pain Inventory will be used to measure interference due to pain. Change in pain intensity measured by Brief Pain Inventory (BPI), which uses a scale of 0 to 10. Higher scores indicate worse pain interference.
Dialysis Symptom Burden | 3, 6 and 12 months
  Dialysis symptom burden and severity will be assessed using the Dialysis Symptom Index (DSI). The total score can range from 0 to 150, with higher scores indicating a greater symptom burden.
Self-Efficacy for Managing Chronic Conditions | 3, 6 and 12 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions Short Form 8A will be used; higher scores indicate greater self-efficacy in managing chronic conditions.
Sleep quality | 3, 6 and 12 months
  PROMIS Sleep Disturbance and sleep duration questions will be asked to assess sleep quality. The scale consists of 6 items with a 5-point response scale. Higher scores indicate greater sleep disturbance.
Post Dialysis fatigue | 3, 6 and 12 months
  Single Item Question asking patients length of time it takes to recover from dialysis treatment will be used to assess post dialysis fatigue. Higher recovery time indicates greater post dialysis fatigue
Anxiety | 3, 6 and 12 months
  The Generalized Anxiety Disorder 7-item (GAD-7) scale will be used to assess severity of anxiety symptoms. Scores range from 0 to 21 with higher scores indicating greater anxiety.
Health related quality of life | 3, 6 and 12 months
  RAND 36-Item Short Form Health Survey (SF-36) will be used to measure health related quality-of-life measures. Scores range from 0 to 100 with higher scores indicating better health status.
Perceived Social Support | 3, 6 and 12 months
  The Multi-Dimensional Scale of Perceived Social Support (MSPSS) will be used to assess patients' perceived level of social support. It is a 12 item measure that uses a 5-point Likert scale with higher scores indicating greater perceived social support.
Adherence to dialysis treatments | 3, 6 and 12 months
  Data on missed dialysis treatments will be recorded from dialysis electronic health record
Hospitalization/ER visits | 3, 6 and 12 months
  Data on hospitalizations and ER visits will be collected from the dialysis electronic health records

OTHER OUTCOMES:
Fatigue Assessment Scale | Every 4 weeks during 12 week intervention
  The Fatigue Assessment Scale (FAS) is scored by summing up the responses to each of its 10 items, where each item is rated on a 5-point Likert scale from "never" (1) to "always" (5), resulting in a total score ranging from 10 (minimal fatigue) to 50 (extreme fatigue) ; higher scores indicate greater fatigue severity.
PROMIS Anxiety SF 8A | Every 4 weeks during 12 week intervention
  The PROMIS Anxiety SF 8A is scored by summing up the responses to each of the 8 questions, where each question is rated on a 5-point scale (1=never to 5=always), resulting in a raw score; this raw score is then converted into a T-score using a reference table to provide a standardized measure of anxiety severity, with a mean T-score of 50 and a standard deviation of 10 across the general population.
PROMIS Depression SF 8A | Every 4 weeks during 12 week intervention
  The PROMIS Depression SF 8A is scored by summing up the responses to each of the 8 questions, where each question is rated on a 5-point scale from 1 ("Never") to 5 ("Always"), resulting in a raw score; this raw score is then converted into a T-score using a provided table to interpret the severity of depression, with higher T-scores indicating greater depression severity.
Visual Analog Scale (VAS) for Pain | Every 4 weeks during 12 week intervention
  A Visual Analog Scale (VAS) for pain is a simple pain measurement tool where a patient marks a point on a 10cm line to indicate the intensity of their pain, with one end representing "no pain" and the other end representing "worst pain imaginable"; the score is determined by measuring the distance from the "no pain" end to the mark made by the patient, usually in centimeters, providing a numerical value representing their pain level

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Jhamb, MD, MPH, Principal Investigator — University of Pittsburgh; Mark L Unruh, MS, MS, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - UNM, Albuquerque, New Mexico
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All subject-level clinical, survey, and laboratory will be preserved and shared. Data will be deidentified before submission.
  The study protocol, date collection forms/case report forms, data dictionary, manual of operations, interview guides, qualitative analysis codebook and a glossary of domain-specific terms will be submitted.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Baseline data (defined as any data collected prior to any intervention), such as demographics, tabular clinical data will be submitted within 4 months after enrollment is completed and released through the repositories 4 months after that. After the study is complete and unblinded, the study team will submit all remaining scientific data to the data repositories and will update the RCT status to "complete" in clinicaltrials.gov. This data will be released 12 months after the end of the study. Under the current repository policies, data will be preserved and available for the wider research community in perpetuity.
Access Criteria: To maximize the appropriate sharing of scientific data and protect research participants' privacy and confidentiality, reuse of this dataset should use the following Data Use Limitations (DULs) under Controlled Access that is made available by a data repository only after approval of the request by the repository's independent review panel process.